CLINICAL TRIAL: NCT06952296
Title: Study of the Effectiveness of Dydrogesterone in the Treatment of Endometriosis-related Pain
Acronym: Daisy
Status: Not yet recruiting | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: DYDR-524-0516
Record Dates: First submitted 2025-04-10; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Dydrogesterone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dydrogesterone group
  Interventions: Drug: Dydrogesterone

INTERVENTIONS:
Drug: Dydrogesterone — The duration of treatment with dydrogesterone is determined by the physician before inclusion in the study and will last for 6 menstrual cycles ("Cycle" used in the protocol refers to menstrual cycle. 1 cycle is 28 days on average)

SUMMARY:
The study is an observational, multicenter, prospective, single arm study to evaluate the efficacy of dydrogesterone in endometriosis-related pain (EAP).

ELIGIBILITY:
Inclusion Criteria:

* Female, ≥18 and ≤45 years of age.
* With normal menstrual cycles (according to the International Federation of Gynecology and Obstetrics [FIGO]-2018 classification system) in the preceding 6 months before Cycle 0, defined as menstrual frequency ≥24 to ≤38 days, menstrual duration ≤8 days, shortest to longest cycle variation ≤7-9 days, normal flow volume (patient determined) and no intermenstrual bleeding.
* Have clinically or surgically diagnosed endometriosis according to routine clinical practice.
* Complaints of ERP.
* Prescribed treatment with Duphaston® according to the local approved label for treatment of endometriosis 10 mg BID or TID from the 5th to the 25th day of the menstrual period.
* Signed informed consent form (ICF).

Exclusion Criteria:

* With definite diagnosis of adenomyosis confirmed by clinical diagnosis or histopathology.
* Routine consumption of analgesics other than for the pain of endometriosis.
* Patients receiving hormonal treatment (e.g., dienogest, levonorgestrel releasing intrauterine system, dydrogesterone, etc.) or hormonal contraceptives (including intrauterine devices, contraceptive patches, contraceptive rings, oral contraceptives, etc.) during the previous menstrual cycle prior to Cycle 0.
* Ongoing pregnancy.
* Menopause or premature ovarian failure.
* Had surgery within 3 months before enrollment or have planned surgery during the study.
* Any coexisting disease(s) with or without chronic concomitant medication that may affect the assessment of pain intensity at the investigator's judgment.
* With any metabolic and genetic diseases that may affect pregnancy and fetus at the investigator's judgment.
* With contraindications for dydrogesterone treatment listed in the locally approved label (instructions for the medical use of Duphaston®).
* Other conditions that made the patient's participation impossible (based on the investigator's decision).
* Fertility treatments requiring assisted reproductive technology.
* Patients simultaneous participating in any interventional clinical study during observation period.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: This study is planned to enroll 250 patients who have endometrosis-related pain (ERP) (dysmenorrhea, Chronic pelvic pain (CPP), dyspereunia, and other ERP) and are planned to be treated with dydrogesterone per the physician's decision.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in visual analogue scale (VAS) score of dysmenorrhea, Chronic Pelvic Pain (CPP), dyspareunia, and other Endometriosis related Pain (ERP) after dydrogesterone treatment from baseline to Cycle 6. | From baseline to Cycle 6 ("Cycle" refers to menstrual cycle, 1 cycle is 28 days on average)
  The VAS consists of a 100-mm line with the end points no pain and worst pain, which "absence of pain" corresponds to the value of "0" and unbearable pain corresponding to the value of "100" . Patients will be asked to point the average pain intensity throughout the last menstrual cycle.

SECONDARY OUTCOMES:
Changes in visual analogue scale (VAS) score of dysmenorrhea, Chronic Pelvic Pain(CPP), dyspareunia, and other Endometriosis related Pain (ERP) after dydrogesterone treatment from baseline to Cycle 3. | From baseline to Cycle 3 ("Cycle" refers to menstrual cycle, 1 cycle is 28 days on average)
  The visual analogue scale (VAS) consists of a 100-mm line with the end points no pain and worst pain, which "absence of pain" corresponds to the value of "0" and unbearable pain corresponding to the value of "100". Patients will be asked to point the average pain intensity throughout the last menstrual cycle.
Changes in Endometriosis Health Profile Questionnaire-30 (EHP-30) after dydrogesterone treatment from baseline to Cycle 3 and Cycle 6. | From baseline to Cycle 3 and Cycle 6 ("Cycle" refers to menstrual cycle, 1 cycle is 28 days on average)
  For the EHP-30, scale scores are standardized on a range from 0 to 100. The higher scores indicate worse health status.
Changes in score of pain domain of Endometriosis Health Profile Questionnaire (EHP-30) from baseline to Cycle 3 and Cycle 6. | From baseline to Cycle 3 and Cycle 6 ("Cycle" refers to menstrual cycle, 1 cycle is 28 days on average)
  For the pain domain of EHP-30, scale scores are standardised on a range from 0 to 100. The higher scores indicate more severe pain.
Changes in sexual well-being after dydrogesterone treatment by 5-points Likert scale from baseline to Cycle 3 and Cycle 6. | From baseline to Cycle 3 and Cycle 6 ("Cycle" refers to menstrual cycle, 1 cycle is 28 days on average)
  A patient-reported sexual wellbeing by 5-points Likert scale proposes patients to rate themselves on a 5-point scale as being "very satisfied, satisfied, ordinarily, rather not satisfied, not satisfied"
Changes in menstrual cycle duration from baseline to Cycle 3 and Cycle 6. | From baseline to Cycle 3 and Cycle 6 ("Cycle" refers to menstrual cycle, 1 cycle is 28 days on average)
The number of days per menstrual cycle when analgesics are taken at baseline, Cycle 3, and Cycle 6. | At baseline, Cycle 3, and Cycle 6 ("Cycle" refers to menstrual cycle, 1 cycle is 28 days on average)
The proportion of participants with amenorrhea, infrequent bleeding, frequent bleeding, irregular bleeding, prolonged bleeding upon treatment with dydrogesterone at baseline, Cycle 3, and Cycle 6. | At baseline, Cycle 3, and Cycle 6 ("Cycle" refers to menstrual cycle, 1 cycle is 28 days on average)
The absolute number and percentage of adverse drug reactions (ADRs) / other pharmacovigilance-relevant information (OPRI) reported with dydrogesterone treatment. | Time Frame: From informed consent to last contact (refers to cycle 6 visit, where "Cycle" refers to menstrual cycle, 1 cycle is 28 days on average) or 5 half-lives (75 hours from the last dose), whichever is longer.